CLINICAL TRIAL: NCT05059860
Title: An Evaluation of the Tandem IQ Insulin Pump and DEXCOM G6 Continuous Glucose Monitoring Hybrid Closed Loop Insulin Delivery System (Control-IQ) on Patient Wellbeing and Diabetes Control in Adults With Type 1 Diabetes
Brief Title: Dexcom Hybrid Closed Loop Insulin Pump Study in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 299847
Record Dates: First submitted 2021-09-08; First posted 2021-09-28 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Tandem Control IQ Hybrid Closed Loop Insulin Delivery System — The Tandem Control IQ hybrid closed loop insulin delivery system is made up of an externally worn Tandem insulin pump which communicates wirelessly to the Dexcom G6 CGM worn as a patch on the skin. The CGM measures glucose levels transmitting them into the computer within the pump. The computer then calculates how much insulin is required then dose delivery completes the cycle. The Control-IQ™ advanced technology adjusts insulin delivery to avoid glycaemic excursions, while still allowing the user to manually bolus at mealtimes.

SUMMARY:
Treatment of Type 1 diabetes requires daily insulin therapy given by either multiple daily injections or by continuous infusion via a pump. The insulin dose is calculated taking into consideration blood glucose levels, food intake and activity levels, aiming to avoid high and low readings.

The Tandem t:slim X2™ insulin pump has recently become available in NHS Scotland and can link with the Dexcom G6 continuous glucose monitoring (CGM) system.

The Tandem Control IQ hybrid closed loop system is made up of the Tandem insulin pump communicating wirelessly with the Dexcom G6 CGM. The algorithm within the pump then automatically controls the background (basal) insulin infusion rate. Manually delivered bolus insulin is still required for meals. This system is designed to finely tune insulin delivery and increase the amount of time that glucose is in the target range, reducing hypoglycaemia and hyperglycaemia.

Insulin pumps are funded by NHS Scotland, but the Dexcom G6 continuous glucose monitoring system is not, so this hybrid closed loop system is not currently routinely available in NHS Scotland.

The purpose of this study is to gain experience of this system and investigate how effective and acceptable the hybrid closed loop system is for people in Scotland. Participants will be provided with the Dexcom G6 CGM device to link to their current pump to create the hybrid closed loop system for the duration of the study.

30 people with Type 1 diabetes who have been using the Tandem pump for at least one month will be invited to participate.

The study will include a screening visit, a 30 day run-in period, 52 week treatment period and 12 week follow-up period. Diabetes control will be measured using HbA1c and downloaded information from the hybrid closed loop system. Participants will also complete questionnaires and a reflective diary.

DETAILED DESCRIPTION:
In those without diabetes insulin is automatically secreted according to requirement. The background insulin secretion rate will vary depending on need, and is affected by many factors e.g. activity or stress levels. When a person eats the rise of glucose is sensed and insulin automatically secreted to keep the glucose within a narrow range.

People with Type 1 diabetes cannot make insulin to control their blood glucose. Insulin is therefore required as treatment. This is given subcutaneously by injection or using an infusion pump. Both background insulin is required and boluses of insulin given when carbohydrate is eaten.

It is difficult to accurately calculate and deliver the correct amount of insulin. More recently standard treatment involved giving one of two injections of long acting insulin and more frequent injections of fast acting insulin when carbohydrate is ingested. The dose of insulin is determined by measuring the ambient glucose level, knowing the amount of carbohydrate in any meal and predicting activity during the subsequent four or five hours.

Insulin pumps can be used to provide a pre-tuned variable background insulin infusion with manual intervention to deliver boluses of insulin with food.

In Scotland many people have now replaced finger prick glucose testing with flash glucose monitoring. This uses a small subcutaneous needle that senses subcutaneous glucose levels and, when scanned this sensor will provide a measure of subcutaneous glucose and information on the last 8 hours of glucose values (Flash Glucose monitoring). This system does not currently link to an insulin pump.

The Tandem insulin pump has recently become available in NHS Scotland for those already established on pump therapy.

The Dexcom G6 continuous glucose monitoring (CGM) system provides continuous glucose monitoring (without requiring any scanning by the patient) but is not currently funded within NHS Scotland, except for special circumstances. This system does communicate via bluetooth with the T-slim insulin pump.

The Tandem Control IQ insulin delivery system uses the link between the dexcom glucose sensor and pump to control the background insulin delivery and has been shown to work well in those studied. Patients still have to administer insulin when ingesting carbohydrate. This system is described as a hybrid closed loop system.

Problems that can potentially occur using this system include loss of communication between sensor and pump (bluetooth or wired connection), the algorithm not working or glucose readings out with the set ranges resulting in the automatic system turning off.

It is also unknown how acceptable the 'loss of control' is to a more general diabetes population as individuals with diabetes are used to making all the insulin dose decisions very frequently across each day. Confidence in these systems, both by patients and clinicians will be vital if these are to be introduced into more general use.

Therefore, the potential for these systems to have a major impact for people with diabetes is clear, but further understanding of the effectiveness and acceptability of such systems in the Scottish population is required.

The Investigator's aim is to investigate the effect of this system compared to current 'best practice' in Scotland, to gain experience in using this system and to investigate the acceptability of this system in the Scottish population.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 1 diabetes
* Established on the Tandem pump for at least 1 month, using novorapid or humalog insulin
* HbA1c 40-90 mmol/mol inclusive within the previous 30 days or taken at screening
* Total daily dose of insulin 10-100 units
* Willing to attend study visits and complete all study assessments
* Able to give informed consent

Exclusion Criteria:

* Pregnant or planning pregnancy
* Any disorder which, in the investigators' opinion might jeopardise the patient's safety or compliance with the protocol
* Life expectancy less than one year
* Severe renal impairment (eGFR <30ml/min)
* Weight <25kg
* Patients prescribed hydroxycarbamide

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 30 patients with Type 1 diabetes will be recruited in NHS Lothian
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
HbA1c | Change from baseline to 20 days after initiation of the sensor, and at 4, 12, 26, 52 and 64 weeks after initiation of the Control-IQ hybrid closed loop system
  Measurement of HbA1c
Severe hypoglycaemia | Change from the 12 weeks before baseline measures to 20 days after initiation of the sensor, and at 4, 12, 26, 52 and 64 weeks after initiation of the Control-IQ hybrid closed loop system.
  Self reported severe hypoglycaemia
Time in range | Change from baseline to 4, 12, 26 and 52 weeks after initiation of the Control-IQ hybrid closed loop system
  Percentage of time glucose is in range (download of Dexcom results)
Time in hypoglycaemia | Change from baseline to 4, 12, 26 and 52 weeks after initiation of the Control-IQ hybrid closed loop system.
  Percentage of time hypoglycaemic
Time Control IQ system not in use | From baseline to 4, 12, 26 and 52 weeks after initiation of the system.
  Time when the Control-IQ hybrid closed loop system is not in use

SECONDARY OUTCOMES:
Diabetes distress score | Change from baseline to 4, 12, 26, 52 and 64 weeks after initiation of the Control-IQ hybrid closed loop system.
  Diabetes distress score. The Diabetes Distress Score yields a total diabetes distress scale score plus 4 sub scale scores, each addressing a different kind of distress. The score is the sum of the patient's responses to the appropriate items divided by the number of items in that scale. A mean question score of 3 or higher (moderate distress) as a level of distress is worthy of clinical attention.
Problem Areas In Diabetes questionnaire | Change from baseline to 4, 12, 26, 52 and 64 weeks after initiation of the Control-IQ hybrid closed loop system.
  Problem Areas In Diabetes questionnaire. Each question has five possible answers with a value from 0 to 4, with 0 representing "no problem" and 4 "a serious problem".
  The scores are added up and multiplied by 1.25, generating a total score between 0 - 100.
  Patients scoring 40 or higher may be at the level of "emotional burnout" and warrant special attention.
  PAID scores in these patients may drop 10-15 points in response to educational and medical interventions.
  An extremely low score (0-10) combined with poor glycaemic control may be indicative for denial
Patient experience diary | Change from baseline to 4, 12, 26, 52 and 64 weeks after initiation of the Control-IQ hybrid closed loop system.
  Patient written report of experience using hybrid closed loop system
Hospital Anxiety and Depression questionnaire | Change from baseline to 4, 12, 26, 52 and 64 weeks after initiation of the Control-IQ hybrid closed loop system.
  Hospital Anxiety and Depression questionnaire. Minimum score is 0, maximum score is 21. 0-7 = Normal, 8-10 = Borderline abnormal (borderline case), 11-21 = Abnormal (case)

OTHER OUTCOMES:
Gold Hypoglycaemia questionnaire | Change from baseline to 4, 12, 26, 52 and 64 weeks after initiation of the Control-IQ hybrid closed loop system.
  Gold hypoglycaemia questionnaire. The Gold score measures hypoglycaemia awareness. Minimum score is 1 - always aware, Maximum score is 7 - never aware. The higher the score the greater the risk of severe hypoglycaemia

CONTACTS AND LOCATIONS:
Overall Officials: John McKnight, Principal Investigator — NHS Lothian
Locations (1):
- Professor John McKnight, Edinburgh, Lothian, United Kingdom